CLINICAL TRIAL: NCT03884426
Title: Genetic and Phenotypic Characteristics of Mitral Valve Prolapse
Acronym: MVP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Collaborators: University Hospital, Brest (Other); Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC12_0143
Record Dates: First submitted 2013-03-21; First posted 2019-03-21 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Mitral Valve Prolapse; Genetic Disease
Keywords: Mitral valve prolapse; genetic; echocardiography
MeSH Terms: conditions — Mitral Valve Prolapse; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with MVP: The patients concerned are patients with known or recently discovered Barlow-type mitral prolapse, whatever the degree of severity.
- Normal relatives: Related healthy patients, for an average of 6 individuals per family

SUMMARY:
Phenotypic characterisation of MVP by echocardiography in families. Identification of genes involved in MVP.

DETAILED DESCRIPTION:
After clinical identification of patients with MVP, doctors organize 1st degree relative familial screening. A comprehensive echocardiography was carried out along with clinical examination. All echo data were stored for off-line analysis by a sonographer in our Core-lab. Blood was sample at the time of echocardiography in adult patients for DNA analyses. Follow-up for mitral valve changes will be performed after 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age
* with typical mitral valve prolapse
* relatives examined during familial screening

Exclusion Criteria:

* Refusal of the patient

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients of both sex of any age with typical mitral valve prolapse and relatives examined during familial screening
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-12 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
MVP defined by a superior displacement of at least 2 mm | At Day 0
  MVP defined by a superior displacement of at least 2 mm

SECONDARY OUTCOMES:
Comprehensive mitral valve apparatus characterization per size of items (leaflets, chordae, annulus) | At Day 0
  Leaflets length ; Chordae length ; Annulus diameter
Comprehensive mitral valve apparatus characterization per other items (papillary muscle, ventricles) | At Day 0
  Papillary muscles aspect ; Right Ventricle function ; Left Ventricle Ejection Fraction
Comprehensive mitral valve apparatus characterization per size of items (ventricle and atrium sizes) | At Day 0
  Left ventricle and atrium sizes ; right ventricle size ; right Atrium size
Comprehensive mitral valve apparatus characterization per size of items | At Day 0
  Leaflets thickness

OTHER OUTCOMES:
Incidence of cardiac or clinical defects associated with MVP | At Day 0 Follow-up will be carried out at 5 and 10 years
  Atrial septal defect, ventricular septal defect, patent ductus arteriosus, tricuspid or aortic valve abnormalities (prolapse, bicuspid AV…), coarctation, ascending aorta aneurysm

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Probst, PU-PH, Principal Investigator — Nantes University Hospital; Hervé Le Marec, PU-PH, Principal Investigator — Nantes University Hospital; Jean-Jacques Schott, DR, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (3):
- France (3):
  - Brest University Hospital, Brest
  - Nantes University Hospital, Nantes
  - Rennes University Hospital, Rennes

REFERENCES:
- [Derived] Huttin O, Girerd N, Jobbe-Duval A, Constant Dit Beaufils AL, Senage T, Filippetti L, Cueff C, Duarte K, Fraix A, Piriou N, Mandry D, Pace N, Le Scouarnec S, Capoulade R, Echivard M, Sellal JM, Marrec M, Beaumont M, Hossu G, Trochu JN, Sadoul N, Marie PY, Guenancia C, Schott JJ, Roussel JC, Serfaty JM, Selton-Suty C, Le Tourneau T. Machine Learning-Based Phenogrouping in MVP Identifies Profiles Associated With Myocardial Fibrosis and Cardiovascular Events. JACC Cardiovasc Imaging. 2023 Oct;16(10):1271-1284. doi: 10.1016/j.jcmg.2023.03.009. Epub 2023 May 17. PMID 37204382